CLINICAL TRIAL: NCT00003884
Title: A Randomized, Double-Blind, Placebo-Controlled, Multicenter Trial to Evaluate the Safety and Efficacy of Zoledronate (4 and 8 mg) Administered Intravenously as an Adjuvant to Anticancer Therapy to Patients With Any Cancer With Bone Metastases Other Than Breast Cancer, Multiple Myeloma or Prostate Cancer
Brief Title: Zoledronate in Treating Patients With Solid Tumors That Have Spread to the Bone
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novartis (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Purpose: Supportive Care
Other Study IDs: CDR0000067052; NOVARTIS-4244603011
Record Dates: First submitted 1999-11-01; First posted 2004-07-22 (Estimated); Last update posted 2013-02-21 (Estimated); Status verified 2013-02

CONDITIONS: Hypercalcemia of Malignancy; Lung Cancer; Metastatic Cancer; Pain; Unspecified Adult Solid Tumor, Protocol Specific
Keywords: hypercalcemia of malignancy; pain; recurrent non-small cell lung cancer; recurrent small cell lung cancer; unspecified adult solid tumor, protocol specific; bone metastases
MeSH Terms: conditions — Humoral Hypercalcemia Of Malignancy; Lung Neoplasms; Neoplasm Metastasis; Pain; Carcinoma, Non-Small-Cell Lung; Small Cell Lung Carcinoma | interventions — Zoledronic Acid

INTERVENTIONS:
Drug: zoledronic acid
Procedure: quality-of-life assessment

SUMMARY:
RATIONALE: Zoledronate may help to relieve some of the symptoms caused by bone metastases. It is not yet known if zoledronate is more effective than no further therapy in relieving symptoms of bone metastases or preventing disease progression.

PURPOSE: Randomized phase III trial to determine the effectiveness of zoledronate in treating patients who have solid tumors that have spread to the bone.

DETAILED DESCRIPTION:
OBJECTIVES: I. Assess the safety and efficacy of zoledronate in patients with any solid tumor cancer with bone metastases other than breast or prostate cancer. II. Assess the efficacy of zoledronate in preventing skeletal-related events including tumor induced hypercalcemia (TIH), time to first occurrence of skeletal-related event or TIH, skeletal morbidity rate, time to progression of bone metastases, overall survival, and time to overall disease progression in these patients. III. Assess the quality of life and pain in these patients on these regimens.

OUTLINE: This is a randomized, double blind, placebo controlled, multicenter study. Patients are stratified into two groups: patients with lung cancer and patients with all other solid tumor cancers. Patients are randomly assigned to receive 1 of the following treatments: Arm I: Patients receive intravenous zoledronate over 5 minutes every 3 weeks for 9 months. Arm II: Patients receive intravenous zoledronate at a higher dose over 5 minutes every 3 weeks for 9 months. Arm III: Patients receive intravenous placebo over 5 minutes every 3 weeks for 9 months. All patients receive oral calcium daily, and an oral multivitamin supplement. Quality of life is assessed prior to therapy, then at months 3, 6, and 9. Patients are followed every 6 months for survival.

PROJECTED ACCRUAL: A total of 600 patients will be accrued for this study within 12 months.

ELIGIBILITY:
DISEASE CHARACTERISTICS: Histologically or cytologically confirmed diagnosis of any cancer other than breast cancer, multiple myeloma, or prostate cancer Objective evidence of bone metastases discovered within 6 weeks of study entry (patients who at screening present with an ECOG score of 2) No study entry restrictions for bone metastases for patients with an ECOG of 0 and 1 No symptomatic brain metastases

PATIENT CHARACTERISTICS: Age: 18 and over Performance status: ECOG 0-2 Life expectancy: Not specified Hematopoietic: Not specified Hepatic: Bilirubin no greater than 2.5 mg/dL for liver metastases Renal: Creatinine no greater than 3.0 mg/dL Calcium at least 8.0 mg/dL but less than 12.0 mg/dL Cardiovascular: No history of severe cardiovascular disease within past 6 months (e.g., congestive heart failure) No hypertension refractory to treatment No symptomatic coronary artery disease Other: Not pregnant or nursing Negative pregnancy test Fertile patients must use effective contraception No history of noncompliance to medical regimen

PRIOR CONCURRENT THERAPY: Biologic therapy: Concurrent biologic response modifier therapies allowed Concurrent marketed cytokine or colony stimulating factor therapies allowed Chemotherapy: Concurrent marketed chemotherapy agents allowed (including open label cooperative trials or for supportive care) Endocrine therapy: Concurrent hormonal agents and steroid therapies allowed Concurrent corticosteroid therapy allowed (for chemotherapy induced nausea/vomiting or spinal compression) Radiotherapy: Concurrent radiotherapy to treat extraskeletal and/or skeletal tumor sites allowed Surgery: Prior surgery to treat or prevent pathological fracture or spinal cord compression allowed Other: At least 30 days since other prior investigational drugs No concurrent bisphosphonate agent At least 30 days since prior bisphosphonate agent (single exposure allowed within prior 12 months)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 600 (Estimated)
Dates: Start 1998-08; Primary Completion 2001-01 (Actual); Study Completion 2001-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Robert Knight, MD, Study Chair — Novartis Pharmaceuticals
Locations (55):
- United States (55):
  - SORRA Research Center, Birmingham, Alabama
  - Brookwood ACCC, Birmingham, Alabama
  - University of Alabama Comprehensive Cancer Center, Birmingham, Alabama
  - Highlands Oncology Group, Springdale, Arkansas
  - Columbia South Valley Hospital, Gilroy, California
  - Pacific Shores Medical Group, Long Beach, California
  - Veterans Affairs Medical Center - West Los Angeles, Los Angeles, California
  - Jonsson Comprehensive Cancer Center, UCLA, Los Angeles, California
  - Southwest Cancer Care, Poway, California
  - Cancer and Blood Institute of the Desert, Rancho Mirage, California
  - Oncology Clinic, P.C., Colorado Springs, Colorado
  - Veterans Affairs Medical Center - Denver, Denver, Colorado
  - Vincent T. Lombardi Cancer Research Center, Georgetown University, Washington D.C., District of Columbia
  - Veterans Affairs Medical Center - Miami, Miami, Florida
  - Oncology-Hematology Group of South Florida, Miami, Florida
  - H. Lee Moffitt Cancer Center and Research Institute, Tampa, Florida
  - American Medical Research Institute, Inc., Atlanta, Georgia
  - Oncology Care Center - Belleville, Belleville, Illinois
  - Fort Wayne Medical Oncology and Hematology, Inc., Fort Wayne, Indiana
  - University of Iowa Hospitals and Clinics, Iowa City, Iowa
  - Louisiana State University Medical Center, Lafayette, Louisiana
  - Ochsner Clinic, New Orleans, Louisiana
  - Louisiana State University Health Sciences Center - Shreveport, Shreveport, Louisiana
  - Maine Center for Cancer Medicine and Blood Disorders, Scarborough, Maine
  - Greater Baltimore Medical Center and Cancer Center, Baltimore, Maryland
  - New England Medical Center Hospital, Boston, Massachusetts
  - New England Hematology/Oncology Associates, P.C., Wellesley, Massachusetts
  - Henry Ford Hospital, Detroit, Michigan
  - Spectrum Health and DeVos Children's Hospital, Grand Rapids, Michigan
  - St. Mary's/Duluth Clinic Health System, Duluth, Minnesota
  - Hubert H. Humphrey Cancer Center, Robbinsdale, Minnesota
  - Kansas City Internal Medicine, Kansas City, Missouri
  - Missouri Baptist Cancer Center, St Louis, Missouri
  - Veterans Affairs Medical Center - Reno, Reno, Nevada
  - Veterans Affairs Medical Center - East Orange, East Orange, New Jersey
  - Brookdale University Hospital and Medical Center, Brooklyn, New York
  - North Shore University Hospital, Manhasset, New York
  - New York Presbyterian Hospital - Cornell Campus, New York, New York
  - University of Rochester Cancer Center, Rochester, New York
  - Albert Einstein Comprehensive Cancer Center, The Bronx, New York
  - Raleigh Internal Medicine, Raleigh, North Carolina
  - Cleveland Clinic Cancer Center, Cleveland, Ohio
  - Hematology Oncology Consultants Inc, Columbus, Ohio
  - University of Oklahoma College of Medicine, Oklahoma City, Oklahoma
  - Regional Cancer Center - Erie, Erie, Pennsylvania
  - Milton S. Hershey Medical Center, Hershey, Pennsylvania
  - University of Pittsburgh Cancer Institute, Pittsburgh, Pennsylvania
  - Palmetto Hematology/Oncology Associates, Spartanburg, South Carolina
  - Dial Research Associates, Brentwood, Tennessee
  - Methodist Hospitals of Memphis, Memphis, Tennessee
  - Cancer Specialist of South Texas. P.A., Corpus Christi, Texas
  - University of Texas Health Center at Tyler, Tyler, Texas
  - Huntsman Cancer Institute, Salt Lake City, Utah
  - Danville Hematology and Oncology, Inc., Danville, Virginia
  - Swedish Cancer Institute, Seattle, Washington